CLINICAL TRIAL: NCT02431052
Title: A Phase 2, Randomized, Double-blind, Vehicle-controlled, Dose-ranging Study of DRM01B Topical Gel in Subjects With Acne Vulgaris
Brief Title: A Dose-ranging Study of DRM01 in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRM01B-ACN02
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Olumacostat Glasaretil Gel, Vehicle QD (Placebo Comparator): Olumacostat Glasaretil Gel, Vehicle, applied once daily to the face for 12 weeks
  Interventions: Other: Vehicle
- Olumacostat Glasaretil Gel, Vehicle BID (Placebo Comparator): Olumacostat Glasaretil Gel, Vehicle, applied twice daily to the face for 12 weeks
  Interventions: Other: Vehicle
- Olumacostat Glasaretil Gel, 4.0% QD (Experimental): Olumacostat Glasaretil Gel, 4.0%, applied once daily to the face for 12 weeks
  Interventions: Drug: Olumacostat Glasaretil
- Olumacostat Glasaretil Gel, 7.5% QD (Experimental): Olumacostat Glasaretil Gel, 7.5%, applied once daily to the face for 12 weeks
  Interventions: Drug: Olumacostat Glasaretil
- Olumacostat Glasaretil Gel, 7.5% BID (Experimental): Olumacostat Glasaretil Gel, 7.5%, applied twice daily to the face for 12 weeks
  Interventions: Drug: Olumacostat Glasaretil

INTERVENTIONS:
Drug: Olumacostat Glasaretil
  Other Names: DRM01B
  Arms: Olumacostat Glasaretil Gel, 4.0% QD; Olumacostat Glasaretil Gel, 7.5% BID; Olumacostat Glasaretil Gel, 7.5% QD
Other: Vehicle
  Arms: Olumacostat Glasaretil Gel, Vehicle BID; Olumacostat Glasaretil Gel, Vehicle QD

SUMMARY:
The objectives of this study are to assess the safety and efficacy DRM01 Topical Gel compared to vehicle in patients with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Male or non-pregnant, non-lactating females.
* Age ≥ 18 years.
* Clinical diagnosis of facial acne vulgaris defined as:
* At least 20 inflammatory lesions
* At least 20 non-inflammatory lesions
* Investigator Global Assessment of 3 or greater.

Exclusion Criteria:

* Active cystic acne or acne conglobata, acne fulminans, and secondary acne.
* Two or more active nodulocystic lesions.
* Screening clinical chemistry or hematology laboratory value that is considered clinically significant, in the opinion of the Investigator.
* Abnormal findings on screening ECG, deemed clinically significant, by the Investigator.
* Subjects who are actively participating in an experimental therapy study or who have received experimental therapy within 30 days or 5 half-lives (whichever is longer) of the Baseline visit.
* Subjects who are a poor medical risk because of other systemic diseases or active uncontrolled infections, in the opinion of the investigator.
* Treatment with over-the-counter topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, α-hydroxy/glycolic acid on the face within 2 weeks prior to Baseline.
* Treatment with systemic corticosteroids (use of intranasal and inhaled corticosteroids allowed for seasonal allergies and asthma) within 4 weeks prior to Baseline.
* Treatment with systemic antibiotics or systemic anti-acne drugs or systemic anti-inflammatory drugs within 4 weeks prior to Baseline.
* Prescription topical retinoid use on the face within 4 weeks of Baseline (e.g., tretinoin, tazarotene, adapalene).
* Treatment with a new hormonal therapy or dose change to existing hormonal therapy within 12 weeks prior to Baseline. Dose and frequency of use of any hormonal therapy started more than 12 weeks prior to Baseline must remain unchanged throughout the study. Hormonal therapies include, but are not limited to, estrogenic and progestational agents such as birth control pills.
* Prior use of androgen receptor blockers (such as spironolactone or flutamide).
* Oral retinoid use (e.g., isotretinoin) within 12 months prior to Baseline or vitamin A supplements greater than 10,000 units/day within 6 months of Baseline.
* Facial procedures (chemical or laser peel, microdermabrasion, etc.) within the past 8 weeks or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Zib, Study Director — Dermira, Inc.
Locations (34):
- United States (28):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - T. Joseph Raoof, MD, Inc., Encino, California
  - University Clinical Trials, Inc., San Diego, California
  - Tory Sullivan MD PA, North Miami Beach, Florida
  - International Clinical Research - US, LLC, Sanford, Florida
  - MOORE Clinical Research, Inc., Tampa, Florida
  - Visions Clinical Research, Wellington, Florida
  - DermResearch, PLLC, Louisville, Kentucky
  - Lawrence J. Green, MD, LLC, Rockville, Maryland
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Las Vegas Dermatology, Las Vegas, Nevada
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Skin Search of Rochester, Inc., Rochester, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - The Skin Wellness Center, Knoxville, Tennessee
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - DermResearch, Inc, Austin, Texas
  - J&S Studies, Inc., College Station, Texas
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - Suzanne Bruce & Associates, PA. The Center for Skin Research, Houston, Texas
  - Suzanne Bruce & Associates, PA. The Center for Skin Research, Katy, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Premier Clinical Research, Spokane, Washington
- Canada (6):
  - Kirk Barber Research, Calgary, Alberta
  - Enverus Medical Research, Surrey, British Columbia
  - Lynderm Research, Markham, Ontario
  - Windsor Clinical Research, Inc., Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermetologique du Quebec Metropolitain (CRDQ), Québec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olumacostat Glasaretil Gel, Vehicle QD | Olumacostat Glasaretil Gel, Vehicle BID | Olumacostat Glasaretil Gel, 4.0% QD | Olumacostat Glasaretil Gel, 7.5% QD | Olumacostat Glasaretil Gel, 7.5% BID
Started | 53 | 50 | 106 | 110 | 101
Completed | 42 | 46 | 94 | 94 | 86
Not Completed | 11 | 4 | 12 | 16 | 15

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Olumacostat Glasaretil Gel, Vehicle QD | Olumacostat Glasaretil Gel, Vehicle BID | Olumacostat Glasaretil Gel, 4.0% QD | Olumacostat Glasaretil Gel, 7.5% QD | Olumacostat Glasaretil Gel, 7.5% BID | Total
Number analyzed (Participants) | 52 | 50 | 106 | 110 | 101 | 419
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 3 | 10 | 15 | 14 | 48
  Between 18 and 65 years | 46 | 47 | 96 | 95 | 87 | 371
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.8 (7.65) | 26.7 (7.04) | 27 (8.13) | 26.4 (7.96) | 25.9 (8.26) | 26.5 (7.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77 | 83 | 79 | 316
  Male | 14 | 11 | 29 | 27 | 22 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 24 | 27 | 32 | 104
  Not Hispanic or Latino | 38 | 41 | 81 | 83 | 68 | 311
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 1 | 0 | 5
  Asian | 1 | 2 | 4 | 6 | 6 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 1 | 0 | 4
  Black or African American | 16 | 12 | 27 | 24 | 20 | 99
  White | 28 | 33 | 69 | 75 | 72 | 277
  More than one race | 4 | 2 | 3 | 3 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 11 | 12 | 25 | 25 | 24 | 97
  United States | 41 | 38 | 81 | 85 | 77 | 322
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type is a scale to numerically classify skin color, defined by the response to ultraviolet (UV) light with the following categories:
  Type I Burns easily, rarely tans Type II Burns easily, tans minimally Type III Burns moderately, tans gradually Type IV Burns minimally, tans well Type V Rarely burns, tans profusely Type VI Never burns, deeply pigmented
  Participants
    Type I | 1 | 2 | 7 | 12 | 5 | 27
    Type II | 9 | 7 | 17 | 23 | 20 | 76
    Type III | 12 | 17 | 26 | 28 | 30 | 113
    Type IV | 15 | 13 | 25 | 22 | 23 | 98
    Type V | 8 | 4 | 9 | 12 | 13 | 46
    Type VI | 7 | 7 | 22 | 13 | 10 | 59

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Change in Acne Lesion Counts (Inflammatory) From Baseline to Week 12
Description: Mean absolute change in acne lesion counts (inflammatory) from baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Deviation); unit: Lesions
Groups:
- Olumacostat Glasaretil Gel, Vehicle QD: Olumacostat Glasaretil Gel, Vehicle, applied once daily to the face for 12 weeks
  Olumacostat Glasaretil
- Olumacostat Glasaretil Gel, Vehicle BID: Olumacostat Glasaretil Gel, Vehicle, applied twice daily to the face for 12 weeks
  Olumacostat Glasaretil
- Olumacostat Glasaretil Gel, 4.0% QD: Olumacostat Glasaretil Gel, 4.0%, applied once daily to the face for 12 weeks
  Olumacostat Glasaretil
- Olumacostat Glasaretil Gel, 7.5% QD: Olumacostat Glasaretil Gel, 7.5%, applied once daily to the face for 12 weeks
  Vehicle
- Olumacostat Glasaretil Gel, 7.5% BID: Olumacostat Glasaretil Gel, 7.5%, applied twice daily to the face for 12 weeks
  Vehicle
Arm/Group | Olumacostat Glasaretil Gel, Vehicle QD | Olumacostat Glasaretil Gel, Vehicle BID | Olumacostat Glasaretil Gel, 4.0% QD | Olumacostat Glasaretil Gel, 7.5% QD | Olumacostat Glasaretil Gel, 7.5% BID
Number analyzed (Participants) | 52 | 50 | 106 | 110 | 101
Lesions | -10.5 (9.79) | -11.0 (9.04) | -14.6 (9.22) | -14.5 (9.49) | -15.0 (9.35)
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, Vehicle QD vs Olumacostat Glasaretil Gel, Vehicle BID vs Olumacostat Glasaretil Gel, 4.0% QD vs Olumacostat Glasaretil Gel, 7.5% QD vs Olumacostat Glasaretil Gel, 7.5% BID; Test type: Other; p = 0.0006, Cochran-Mantel-Haenszel; ANCOVA with factors of treatment group (combined vehicle as one group) and baseline count as covariate

2. Primary Outcome: Mean Absolute Change in Acne Lesion Counts (Non-inflammatory) From Baseline to Week 12
Description: Mean absolute change in acne lesion counts (non-inflammatory) from baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent-To-Treat
Measure: Least Squares Mean (Standard Deviation); unit: Lesions
Arm/Group | Olumacostat Glasaretil Gel, Vehicle QD | Olumacostat Glasaretil Gel, Vehicle BID | Olumacostat Glasaretil Gel, 4.0% QD | Olumacostat Glasaretil Gel, 7.5% QD | Olumacostat Glasaretil Gel, 7.5% BID
Number analyzed (Participants) | 52 | 50 | 106 | 110 | 101
Lesions | -9.3 (15.62) | -9.3 (15.07) | -15.3 (15.17) | -13.4 (15.42) | -17.5 (15.15)
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, Vehicle QD vs Olumacostat Glasaretil Gel, Vehicle BID vs Olumacostat Glasaretil Gel, 4.0% QD vs Olumacostat Glasaretil Gel, 7.5% QD vs Olumacostat Glasaretil Gel, 7.5% BID; Test type: Other; p = 0.0002, Cochran-Mantel-Haenszel; ANCOVA with factors of treatment group (combined vehicle as one group) and baseline count as covariate

3. Primary Outcome: Percentage of Subjects Who Achieved ≥ 2-grade Improvement and a Grade of 0 or 1 in the Investigator Global Assessment of Acne (IGA) From Baseline to Week 12
Description: Percentage of subjects who achieved ≥ 2-grade improvement and a grade of 0 or 1 in the investigator global assessment of acne (IGA) from baseline to Week 12
  Scoring Criteria for Investigator Global Assessment 0 - Clear skin with no inflammatory or noninflammatory lesions
  1. - Almost clear; rare noninflammatory lesions with no more than one small inflammatory lesion
  2. - Mild severity; greater than Grade 1; some noninflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions)
  3. - Moderate severity; greater than Grade 2; up to many noninflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion
  4. - Severe; greater than Grade 3; up to many noninflammatory and inflammatory lesions, but no more than a few nodular lesions
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Olumacostat Glasaretil Gel, Vehicle QD | Olumacostat Glasaretil Gel, Vehicle BID | Olumacostat Glasaretil Gel, 4.0% QD | Olumacostat Glasaretil Gel, 7.5% QD | Olumacostat Glasaretil Gel, 7.5% BID
Number analyzed (Participants) | 52 | 50 | 106 | 110 | 101
Participants
  Success | 4 | 6 | 23 | 21 | 26
  Failure | 48 | 44 | 83 | 89 | 75
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, Vehicle QD vs Olumacostat Glasaretil Gel, Vehicle BID vs Olumacostat Glasaretil Gel, 4.0% QD vs Olumacostat Glasaretil Gel, 7.5% QD vs Olumacostat Glasaretil Gel, 7.5% BID; Test type: Other; p = 0.0055, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test (vehicle treatment groups included as single combined treatment group)

ADVERSE EVENTS:
Time Frame: Baseline to Week 12
Description: The Total Participants at risk are based on the Safety Population defined as Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Olumacostat Glasaretil Gel, Vehicle QD | Olumacostat Glasaretil Gel, Vehicle BID | Olumacostat Glasaretil Gel, 4.0% QD | Olumacostat Glasaretil Gel, 7.5% QD | Olumacostat Glasaretil Gel, 7.5% BID
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50 | 0/106 | 0/109 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50 | 0/106 | 1/109 | 0/101
Other Adverse Events (participants affected / at risk) | 0/52 | 0/50 | 4/106 | 6/109 | 7/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, Vehicle QD (N=52) | Olumacostat Glasaretil Gel, Vehicle BID (N=50) | Olumacostat Glasaretil Gel, 4.0% QD (N=106) | Olumacostat Glasaretil Gel, 7.5% QD (N=109) | Olumacostat Glasaretil Gel, 7.5% BID (N=101)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, Vehicle QD (N=52) | Olumacostat Glasaretil Gel, Vehicle BID (N=50) | Olumacostat Glasaretil Gel, 4.0% QD (N=106) | Olumacostat Glasaretil Gel, 7.5% QD (N=109) | Olumacostat Glasaretil Gel, 7.5% BID (N=101)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 4 | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes